CLINICAL TRIAL: NCT00497458
Title: Phase II Study of Testosterone Replacement in Women Experiencing Aromatase Inhibitor Side-Effects in Adjuvant Therapy for Breast Cancer
Brief Title: Androgen Therapy for Breast Cancer Patients With Aromatase Inhibitor Induced Side-Effects
Acronym: ART2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Havah Therapeutics Pty Ltd (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Stephen Birrell, Director
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ART2
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer; Arthralgia; Osteoporosis
Keywords: breast; neoplasms; anastrazole; testosterone
MeSH Terms: conditions — Breast Neoplasms; Arthralgia; Osteoporosis; Neoplasms | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arimidex (Placebo Comparator): Arimidex 1 mg plus placebo
  Interventions: Drug: Testosterone
- Arimidex test 40mg (Active Comparator): Arimidex 1mg and testosterone 40mg
  Interventions: Drug: Testosterone
- Arimidex plus test 80mg (Active Comparator): Arimidex 1mg and testosterone 80mg
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — testosterone 40 or 80 mg once a day

SUMMARY:
The purpose of this study is to evaluate whether increasing blood levels of androgen can reduce some of the side-effects of anti-estrogen therapy (Arimidex)

DETAILED DESCRIPTION:
Anastrozole (Arimidex®) is a selective aromatase inhibitor (a drug that interferes with the making of oestrogens). Reduction in serum oestrogen levels in a hormone-receptor positive breast cancer patient is clearly beneficial in delaying the regrowth of breast cancer cells in the body. Anastrozole is effective in reducing serum oestrogen levels which results in several significant side-effects with 2 being of significant importance; joint pain and stiffness and bone thinning or osteoporosis. The question being asked in this trial is if replacement of testosterone to women receiving Anastrozole can have a reduction in these 2 common side-effects. Women normally have circulating in their blood 3 major sex hormones: oestrogen, testosterone and progesterone. Each of these is produced by the ovaries. Oestrogen is also made throughout the body but particularly in body fat. Testosterone can also be made in other parts of the body from hormones (DHEA and DHEAS) that are produced by the adrenal glands. At the time of natural menopause, surgical removal of the ovaries or destruction of the ovaries by chemotherapy, oestrogen and progesterone levels fall precipitously. Testosterone levels however fall more gradually with increasing age such that a woman in her forties has on average only half of the testosterone circulating in her bloodstream as does a woman in her twenties. After a woman has her ovaries removed by surgery or destroyed by chemotherapy testosterone levels can fall by up to fifty percent. However testosterone does not change across menopause, although this varies somewhat between women. Testosterone is known to have many physiological roles in women. Firstly, oestrogen is actually made from testosterone, and without the ability of our bodies to make testosterone we cannot make oestrogen. Testosterone appears to have direct independent effects in different parts of the body, and some women may experience a variety of physical symptoms when their blood levels fall. Anastrazole almost completely blocks the formation of oestrogen from testosterone. Thus the question being asked in this trial is, can increasing the blood level of testosterone reduce specific side-effects caused by reduction availability of hormones in joints and bones.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Undergone a total mastectomy, a lumpectomy or a quadrantectomy for primary breast cancer +/-chemo, +/-radiotherapy
* Have commenced anastrozole therapy within the previous 6 months
* Presence of node negative or positive disease
* Receptor-positive tumors, defined as ER ≥10% of the tumor cells positive by immunocytochemical evaluation
* Postmenopausal whether induced by surgery, radiotherapy (chemotherapy-induced amenorrhea may be difficult to determine they may be amenorrhoeic but still have functioning ovaries), or by being naturally amenorrhoeic, for 1 year or more if younger than 50 and for 6 months if 50 or older
* Postmenopausal levels of FSH/LH/E2 (follicle stimulating hormone, luteinizing hormone, oestrogen) according to the definition of "postmenopausal range" for the laboratory involved
* Have developed arthralgia and associated joint symptoms whilst being treated with anastrozole with a score of 40mm or greater on a pain and stiffness 100mm VAS
* WBC ≥ 3.0 x 109/L, granulocytes ≥ 1.5 X 109/L and platelets ≥ 100 x 109/L.
* AST/SGOT or ALT/SGPT ≤ 3 times ULN Serum creatinine ≤ 2 times ULN

Exclusion Criteria:

* Presence of metastatic disease
* Diabetes mellitus or glucose intolerance defined as a fasting glucose >6mmol/l
* Previous or concomitant other (non-breast cancer) malignancy within the previous 5 years
* Presence of other non-malignant systemic diseases which may prevent prolonged follow-up
* History of coronary artery disease or no history of previous coronary heart disease but at least two other coronary heart disease risk factors: LDL ≥8.8 mg/dL OR if fewer than two other coronary heart disease risk factors: LDL ≥10.45 mg/dL or total fasting cholesterol ≥ 13.2 mg/dL
* Patients on hormone replacement therapy (HRT) within 4 weeks before trial treatment was initiated
* Patients on breast cancer chemoprevention with anti-oestrogens if less than 18 months between stopping and diagnosis of breast cancer
* Are at risk of transmitting Human Immunodeficiency Virus or viral hepatitis via infected blood
* Known hypersensitivity to any component of testosterone
* Unable to comply with study requirements
* Taking the following concomitant medications at the screening visit-bisphosphonate, anti-cancer treatment other than anastrozole (this includes Herceptin).
* Prolonged systemic corticosteroid treatment, except for topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intra-articular). Note: Short duration (< 2 weeks) of systemic corticosteroids is allowed (e.g. for Chronic Obstructive Pulmonary Disease) but not within 1 month prior to randomisation.
* Any investigational drugs
* Systemic hormone replacement therapy
* Pregnant or lactating women
* Patients with history of fragility fracture or low BMD, osteoporosis or osteopenia
* Known liver disease

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Reduces arthralgia and associated joint symptoms as indicated by the change in hand or large joint pain from baseline to 3 months using a 100mm visual analogue scale for pain. | 3 months
Has acceptable safety and tolerability profile with particular reference to androgenic adverse events including acne, hirsutism, and alopecia. | 3 months

SECONDARY OUTCOMES:
Impacts the bone resorption marker CTx | 3 months
Impacts serum HDL, LDL Trg, total Chol, | 3 months
Impacts serum levels of oestrogens, androgens and SHBG levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Birrell, MD PhD, Study Director — Havah Therapeutics Pty Ltd
Locations (1):
- Burnside Breast Centre, Adelaide, South Australia, Australia